CLINICAL TRIAL: NCT03524924
Title: Edoxaban Performance in Senior Citizen With Non-valvular Atrial Fibrillation Evaluated Per Frailty
Brief Title: Edoxaban and Frailty in Senior Individuals
Acronym: ESCAPE
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Vittorio Pengo, Associate Professor, University of Padova
Other Study IDs: 4291/AO/17
Record Dates: First submitted 2018-04-26; First posted 2018-05-15 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; elderly; edoxaban; frailty; SHARE-FI; Stroke; Major bleeding
MeSH Terms: conditions — Atrial Fibrillation; Frailty; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non-frail: Survey of Health, Ageing and Retirement in Europe Frailty Instrument (SHARE-FI) score Female: < 0.3151361243 Male: < 1.211878526
- pre-frail: Survey of Health, Ageing and Retirement in Europe Frailty Instrument (SHARE-FI) score Female: 0.3151361243 to < 2.1301121973 Male: 1.211878526 to < 3.0052612772
- frail: Survey of Health, Ageing and Retirement in Europe Frailty Instrument (SHARE-FI) score Female: 2.1301121973 to < 6 Male: 3.0052612772 to < 7

SUMMARY:
Edoxaban, has shown in clinical registration trials a significant reduction of major bleeding compared to warfarin, especially in elderly patients. Efficacy and safety of edoxaban will be assessed in a cohort of very elderly patients (≥80 years of age) with NVAF. A secondary analysis will correlate outcomes with frailty defined according to SHARE-FI (not-frail, pre-frail or frail).

DETAILED DESCRIPTION:
Aim of the study To assess the efficacy and safety of edoxaban in a cohort of very elderly patients (≥80 years of age) with NVAF.

Edoxaban has never been tested in elderly frail patients. In both sexes, there is a non-linear association between age and frailty. A secondary analysis according to frailty assessment (not-frail, pre-frail or frail) will be also performed.

Study Design Observational prospective cohort study including patients of ≥80 years of age with a new diagnosis of NVAF. Edoxaban 60 mg (or 30 mg for patients with CrCL 15 - 50 mL/min or with body weight ≤ 60 kg) will be administered to all patients. All participants will be stratified according to frailty, as assessed by SHARE-FI score, to non-frail, pre-frail, and frail.

Study Population Patients of both sexes, of ≥80 years of age with a new diagnosis of non-valvular atrial fibrillation and without contraindications to Edoxaban.

Outcomes

The following events will be included as outcomes:

* arterial ischemic events (TIA or stroke documented a CT scan; documented systemic embolism)
* major bleeding events (according to the ISTH definition)
* clinically relevant non-major bleeding (CRNM), defined as bleeding that did not meet the definition of major bleeding, but considered clinically significant (including spontaneous gastrointestinal bleeding or rectal bleeding; macroscopic haematuria or urethral bleeding requiring medical attention; skin haematoma >25 cm2; and gingival bleeding or spontaneous ear-nose-throat bleeding lasting ≥5 min) and/or resulted in discontinuation of study medication18.
* death (divided into cardiovascular death, fatal bleeding and other causes of death).

Follow up Follow-up visits will be performed at 3, 6, 12 and 24 months to assess adherence and compliance to therapy, evaluation of relevant blood test and clinical assessment.

Temporary discontinuation of edoxaban for a planned surgical intervention will be allowed.

Patients will be followed until the occurrence of a first outcome event, permanent discontinuation of edoxaban or the end of follow-up period, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* NVAF diagnosed in the past 30 days
* Age at baseline of 80 years or older with indication for anticoagulation treatment with edoxaban

Exclusion Criteria:

* NVAF diagnosed more than 30 days prior to baseline visit
* Other OAT, except for warfarin or LMWH, already started at the time of baseline visit
* Patients with end stage renal disease (ESRD) (CrCL < 15 mL/min) or on dialysis
* Severe hepatic impairment (defined as Child-Pugh Class B or C or increase in transaminases more than three times the upper reference value of normality) or hepatic disease associated with coagulopathy
* Elevated liver enzymes (ALT/AST > 2 x ULN) or total bilirubin ≥ 1.5 x ULN at baseline
* Recent (within 1 month) or persisting gastrointestinal ulceration
* Active neoplasm
* Known or suspected oesophageal varices
* Arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities
* Life expectancy <1 year
* Concomitant use of strong P-gp drugs which contraindicate edoxaban use12 (e.g. HIV protease inhibitors)
* Clinically significant active bleeding or high risk of bleeding conditions such as: recent brain or spinal injury; recent brain, spinal or ophthalmic surgery; recent intracranial haemorrhage
* Known contraindications or hypersensitivity to the active substance or to any of the excipients of Lixiana
* Lack of acquisition of informed consent or refusal to participate by the subject or family representative

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This is an observational prospective cohort study including patients with a new diagnosis of NVAF.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of arterial ischemic events, major bleeding, and clinically relevant non-major bleeding | Through study completion, an average of 24 months
  Cumulative incidence of arterial ischemic events (stroke/TIA and systemic embolism), major bleeding according to ISTH definition, and clinically relevant non-major bleeding (bleeding not meeting major bleeding criteria but considered clinically significant).
Death | Through study completion, an average of 24 months
  Divided into cardiovascular death, fatal bleeding and other causes of death

SECONDARY OUTCOMES:
Correlation of frailty, as measured with Survey of Health, Ageing and Retirement in Europe - Frailty Instrument, with the cumulative incidence of stroke/TIA, systemic embolism, major bleeding and clinically relevant non-major bleeding. | 24 months
  Patients will be divided into 3 groups according to frailty measured with Survey of Health, Ageing and Retirement in Europe - Frailty Instrument (SHARE-FI) which provides 3 patient categories (non-frail, pre-frail and frail).
  A score of < 0.3151361243 defines non frail female patients; a score of 0.3151361243 to 2.1301121973 defines pre-frail female patients; a score of 2.1301121973 to 6 defines frail female patients.
  A score of < 1.211878526 defines non frail male patients; a score of 1.211878526 to 3.0052612772 defines pre-frail male patients; a score of 3.0052612772 to 7 defines frail male patients.
  Further SHARE-FI score details and calculations are available at: https://sites.google.com/a/tcd.ie/share-frailty-instrument-calculators/.
  Outcome events will be compared among the three groups.
Death | Through study completion, an average of 24 months
  All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Pengo, Prof, Principal Investigator — Padua University Hospital
Locations (1):
- Padua University Hospital, Padua, Italy

REFERENCES:
- [Derived] Denas G, Zoppellaro G, Granziera S, Pagliani L, Noventa F, Iliceto S, Pengo V. Very Elderly Patients With Atrial Fibrillation Treated With Edoxaban: Impact of Frailty on Outcomes. JACC Adv. 2023 Aug 24;2(7):100569. doi: 10.1016/j.jacadv.2023.100569. eCollection 2023 Sep. PMID 38939480